CLINICAL TRIAL: NCT01393964
Title: PH Ib Study of Elotuzumab in Combination With Lenalidomide and Dexamethasone in Subjects With Multiple Myeloma and Normal Renal Function, Severe Renal Impairment, or End Stage Renal Disease Requiring Dialysis
Brief Title: Study of Elotuzumab in Combination With Lenalidomide and Dexamethasone in Subjects With Multiple Myeloma and Various Levels of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-007
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Lenalidomide + Dexamethasone +Elotuzumab (Experimental): Severe Renal Impairment
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Biological: Elotuzumab (BMS-901608; HuLuc63)
- Arm 2: Lenalidomide + Dexamethasone +Elotuzumab (Experimental): End-stage renal disease
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Biological: Elotuzumab (BMS-901608; HuLuc63)
- Arm 3: Lenalidomide + Dexamethasone +Elotuzumab (Experimental): Normal renal function
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Biological: Elotuzumab (BMS-901608; HuLuc63)

INTERVENTIONS:
Drug: Lenalidomide — Capsules, Oral, 15 mg, One capsule every 48 hours through Days 1-21 (Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Revlimid®
Drug: Dexamethasone — Tablets, Oral, 28 mg weekly, on day 1 (cycle 1); days 1, 8, 15, 22 (cycles 2-3; days 1 &15 (cycle 4 and beyond) Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak® Taperpak®
Drug: Dexamethasone — Tablets, Oral, 40 mg, weekly, on days 8, 15 & 22 (cycle 1); days 8 &22 (cycle 4 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak® Taperpak®
Drug: Dexamethasone — Solution, Intravenous, 8 mg, weekly, on day 1 (cycle 1); days 1, 8, 15, 22 (cycles 2-3; days 1 &15 (cycle 4 and beyond) Repeat every 28 days until subject meets criteria for discontinuation of study drug
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak® Taperpak®
Biological: Elotuzumab (BMS-901608; HuLuc63) — Solution, Intravenous, 10 mg/kg, weekly, on day 1 (cycle 1); days 1, 8, 15, 22 (cycles 2-3; days 1 &15 (cycle 4 and beyond), Repeat every 28 days until subject meets criteria for discontinuation of study drug

SUMMARY:
The purpose of the study is to assess the concentration of Elotuzumab in Myeloma patients with very low kidney function including patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Multiple Myeloma (MM) and renal function fitting one of three categories:

  1. Severe renal impairment: estimated creatinine clearance (CrCl) <30 ml/min, but not requiring dialysis
  2. End-stage renal disease: requiring hemodialysis
  3. Normal renal function: estimated CrCl ≥90 ml/min
* Documented evidence of symptomatic MM, either newly diagnosed or relapsed/refractory
* Prior Lenalidomide exposure is permitted only if the subject did not discontinue Lenalidomide due to a Grade ≥3 related Adverse Event (AE)

Exclusion Criteria:

* Monoclonal Gammopathy of Undetermined Significance (MGUS), Waldenstrom's macroglobulinemia, or smoldering myeloma
* Active plasma cell leukemia
* All adverse events of any prior chemotherapy, surgery, or radiotherapy not resolved
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-01-06 (Actual); Primary Completion 2014-03-21 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Investigative Clinical Research Of Indiana, Llc, Indianapolis, Indiana
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - University Of Maryland, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Tennessee Oncology, Pllc, Nashville, Tennessee
  - The University Of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Va Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants were enrolled; 9 did not enter into the treatment period. Reasons for not entering treatment period: 8 no longer met criteria, 1 other.
Groups:
- Elotuzumab + LD in Normal Renal Function(NRF) Participants: Combination of lenalidomide and dexamethasone (LD). Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly (Days 1, 8, 15, 22) for Cycles 2 and 3, and every 2 weeks (Q2W) beginning with Cycle 4 and thereafter until disease progression, discontinuation due to unacceptable toxicity, or other protocol-specified reasons. Lenalidomide dosing was based on creatinine clearance (CrCl) calculated using the Cockcroft-Gault (C-G) formula based on Day 1 creatinine and Day 1 weight measured at each cycle (per product label). Dexamethasone was administered weekly as a 40mg oral dose (po) on weeks without elotuzumab; and as a split dose of 28 mg po 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G Creatinine Clearance CrCl Method was used to determine renal function. NRF = CrCl ≥ 90 milliliters per minute (mL/min).
- Elotuzumab + LD in Severe Renal Impairment(SRI) Participants: Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg IV was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and Q2W beginning with Cycle 4 and thereafter until disease progression, discontinuation due to unacceptable toxicity, or other protocol-specified reasons. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle(per product label). Dexamethasone was administered weekly PO as 40mg dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. SRI = estimated CrCl < 30 ml/min but no dialysis.
- Elotuzumab + LD in End Stage Renal Disease(ESRD) Participants: Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, Q2W beginning with Cycle 4 and thereafter until disease progression, discontinuation due to unacceptable toxicity, or other protocol-specified reasons. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle(per product label). Dexamethasone was administered weekly as a 40mg PO dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. ESRD = requires hemodialysis.
Period: Overall Study
Arm/Group | Elotuzumab + LD in Normal Renal Function(NRF) Participants | Elotuzumab + LD in Severe Renal Impairment(SRI) Participants | Elotuzumab + LD in End Stage Renal Disease(ESRD) Participants
Started | 8 | 9 | 9
Completed | 0 (Completed=treatment on-going) | 0 (Completed=treatment on-going) | 0 (Completed=treatment on-going)
Not Completed | 8 | 9 | 9
Not completed — Disease Progression | 4 | 3 | 5
Not completed — Study drug toxicity | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse event unrelated to study drug | 0 | 3 | 0
Not completed — Subject request stop study treatment | 0 | 1 | 0
Not completed — Subject decided to move to transplant | 1 | 0 | 0
Not completed — Subject switched to commercial supply | 1 | 0 | 2
Not completed — Subject plateaued in terms of effect | 1 | 0 | 0
Not completed — Investigator removed subject from study | 0 | 1 | 0
Not completed — Subject converted to roll-over study | 0 | 1 | 0
Not completed — Subject to receive non-protocol therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug (Treated Population).
Groups:
- Elotuzumab + LD in Normal Renal Function (NRF) Participants: Treatment was administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and every 2 weeks (Q2W) beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on creatinine clearance (CrCl) calculated using the Cockcroft-Gault (C-G) formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg oral dose (po) on weeks without elotuzumab; and as a split dose of 28 mg po 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G Creatinine Clearance CrCl Method was used to determine renal function. NRF =CrCl ≥ 90 milliliters per minute (mL/min).
- Elotuzumab + LD in Severe Renal Impairment (SRI) Participants: Treatment was administered in 28 day cycles: Elotuzumab 10 mg/kg IV was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and Q2W beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly PO as 40mg dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. SRI= estimated CrCl < 30 ml/min but no dialysis.
- Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants: Treatment was administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, Q2W beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg PO dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. ESRD= requires hemodialysis.
- Total: Total of all reporting groups
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants | Total
Number analyzed (Participants) | 8 | 9 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (8.05) | 75.9 (7.70) | 55.6 (11.70) | 63.3 (13.02)
Age, Customized [Number; unit: participants]
  < 65 years | 7 | 1 | 8 | 16
  >=65 and < 75 years | 1 | 3 | 0 | 4
  >= 75 years | 0 | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 5 | 6 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Maximum Observed Serum Concentration (Cmax) of Elotuzumab Following Cycle 1, Day 1 Dose Administration - Grouping by Cockcroft-Gault Creatinine Clearance Method
Description: The quantification of elotuzumab in human serum was performed using a validated Enzyme-linked immunoassay (ELISA). Cycle 1, day 1 sample times for all participants: 0 hour (h) pre-dose, end of infusion, 30 minutes (min) post end of infusion, 2 h, 4 h , and 24 h post end of infusion. Trough samples were obtained in subsequent cycles and at 30 day and 60 day follow-up visits at end of treatment. ESRD had 2 additional samples: immediately prior to and immediately after dialysis. Cmax was measured in micrograms per milliliter (µg/mL). Pharmacokinetic (PK) parameter renal function group assignment criteria differed slightly from the criteria for safety and efficacy analyses (specifically for the SRI group). PK criteria: All participants with at least one pretreatment value ≥ 90 mL/min were assigned to the NRF group. All those with at least one pretreatment value < 30 mL/min were assigned to the SRI group. All those with a screening diagnosis of ESRD, were assigned to the ESRD group.
Time Frame: Day 1 of Cycle 1 to 28 days post dose
Population: The analyses of primary endpoint of PK parameters were conducted by renal functions as determined by CrCl C-G method in those participants who were treated with at least one dose of study drug and had evaluable pre- and post-treatment values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Elotuzumab + LD in Normal Renal Function (NRF) Participants: LD=Combination of lenalidomide and dexamethasone. Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and every 2 weeks (Q2W) beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on creatinine clearance (CrCl) calculated using the Cockcroft-Gault (C-G) formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg oral dose (po) on weeks without elotuzumab; and as a split dose of 28 mg po 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G Creatinine Clearance CrCl Method was used to determine renal function. NRF =CrCl ≥ 90 milliliters per minute (mL/min).
- Elotuzumab + LD in Severe Renal Impairment (SRI) Participants: Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg IV was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and Q2W beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly PO as 40mg dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. SRI= estimated CrCl < 30 ml/min but no dialysis.
- Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants: Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, Q2W beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg PO dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. ESRD= requires hemodialysis.
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 7 | 8
µg/mL | 217 (24) | 226 (10) | 218 (21)
Statistical Analysis 1: Comparison: Elotuzumab + LD in Normal Renal Function (NRF) Participants vs Elotuzumab + LD in Severe Renal Impairment (SRI) Participants; The reference arm is NRF participants; Test type: Superiority or Other; p = 0.704, ANOVA; Ratio of Adjusted Means = 104.096, 90% CI 2-sided [86.983 to 124.576]
Statistical Analysis 2: Comparison: Elotuzumab + LD in Normal Renal Function (NRF) Participants vs Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants; The reference arm is NRF participants; Test type: Superiority or Other; p = 0.965, ANOVA; ratio of adjusted means = 100.454, 90% CI 2-sided [84.453 to 119.488]

2. Primary Outcome: Geometric Mean Area Under Serum Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration AUC(0-T) and From Time Zero Extrapolated to Infinite Time AUC(INF) of Elotuzumab Following Cycle 1, Day 1 - Grouping by C-G CrCl Method
Description: The quantification of elotuzumab in human serum was performed using validated ELISA. Cycle 1, day 1 sample times for all participants: 0 hour (h) pre-dose, end of infusion, 30 minutes (min) post end of infusion, 2 h, 4 h , and 24 h post end of infusion. Trough samples were obtained in subsequent cycles and at 30 day and 60 day follow-up visits at end of treatment. ESRD participants had 2 additional sample times: immediately prior to and immediately after dialysis. AUC was measured in µg*h/mL. PK parameter renal function group assignment criteria differed slightly from the criteria for safety and efficacy analyses (specifically for the SRI group). PK criteria: All participants with at least one pretreatment value ≥ 90 mL/min were assigned to the NRF group. All those with at least one pretreatment value < 30 mL/min were assigned to the SRI group. All those with a screening diagnosis of ESRD, were assigned to the ESRD group
Time Frame: Day 1 of Cycle 1 to 28 days post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Groups:
- Elotuzumab + LD in Normal Renal Function (NRF) Participants: LD=Combination of lenalidomide and dexamethasone. Treatment was administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and every 2 weeks (Q2W) beginning with Cycle 4 and thereafter. Lenalidomide dosing was based on creatinine clearance (CrCl) calculated using the Cockcroft-Gault (C-G) formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg oral dose (po) on weeks without elotuzumab; and as a split dose of 28 mg po 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G Creatinine Clearance CrCl Method was used to determine renal function. NRF =CrCl ≥ 90 milliliters per minute (mL/min).
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 7 | 8
µg*h/mL
  AUC (0-T) | 39559 (28) | 50080 (20) | 45937 (31)
  AUC (INF) | 46401 (39) | 60255 (31) | 51227 (39)
Statistical Analysis 1: Comparison: Elotuzumab + LD in Normal Renal Function (NRF) Participants vs Elotuzumab + LD in Severe Renal Impairment (SRI) Participants; AUC(0-T). The reference arm is NRF participants; Test type: Superiority or Other; p = 0.164, ANOVA; Ratio of Adjusted Means = 126.596, 90% CI 2-sided [95.52 to 167.783]
Statistical Analysis 2: Comparison: Elotuzumab + LD in Normal Renal Function (NRF) Participants vs Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants; AUC(0-T). The reference arm is NRF participants; Test type: Superiority or Other; p = 0.355, ANOVA; Ratio of Adjusted Means = 116.123, 90% CI 2-sided [88.458 to 152.439]
Statistical Analysis 3: Comparison: Elotuzumab + LD in Normal Renal Function (NRF) Participants vs Elotuzumab + LD in Severe Renal Impairment (SRI) Participants; AUC (INF). The reference arm is NRF participants; Test type: Superiority or Other; p = 0.228, ANOVA; Ratio of Adjusted Means = 129.858, 90% CI 2-sided [90.366 to 186.609]
Statistical Analysis 4: Comparison: Elotuzumab + LD in Normal Renal Function (NRF) Participants vs Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants; AUC(INF). The reference arm is NRF participants; Test type: Superiority or Other; p = 0.642, ANOVA; Ratio of Adjusted Means = 110.400, 90% CI 2-sided [76.825 to 158.647]

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Who Died
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: From first dose (Day 1) to last dose plus 60 days (Assessed up to July 2016, approximately 54 months)
Population: All participants who received at least one dose of study treatment (at least one dose of any drug) were summarized.
Measure: Number; unit: participants
Groups:
- Elotuzumab + LD in Normal Renal Function (NRF) Participants: LD=Combination of lenalidomide and dexamethasone. Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly (Days 1, 8, 15, 22) for Cycles 2 and 3, and every 2 weeks (Q2W) beginning with Cycle 4 and thereafter until disease progression, discontinuation due to unacceptable toxicity, or other protocol-specified reasons. Lenalidomide dosing was based on creatinine clearance (CrCl) calculated using the Cockcroft-Gault (C-G) formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg oral dose (po) on weeks without elotuzumab; and as a split dose of 28 mg po 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G Creatinine Clearance CrCl Method was used to determine renal function. NRF =CrCl ≥ 90 milliliters per minute (mL/min).
- Elotuzumab + LD in Severe Renal Impairment (SRI) Participants: Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg IV was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, and Q2W beginning with Cycle 4 and thereafter until disease progression, discontinuation due to unacceptable toxicity, or other protocol-specified reasons. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly PO as 40mg dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. SRI= estimated CrCl < 30 ml/min but no dialysis.
- Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants: Elotuzumab + LD were administered in 28 day cycles: Elotuzumab 10 mg/kg intravenous (IV) was administered on Day 1 only for Cycle 1, weekly for Cycles 2 and 3, Q2W beginning with Cycle 4 and thereafter until disease progression, discontinuation due to unacceptable toxicity, or other protocol-specified reasons. Lenalidomide dosing was based on CrCl calculated using the C-G formula based on Day 1 creatinine and Day 1 weight measured at each cycle. Dexamethasone was administered weekly as a 40mg PO dose on weeks without elotuzumab; and as a split dose of 28 mg PO 3 to 24 hours before and 8 mg IV at least 45 minutes before the start of the elotuzumab infusion on weeks with elotuzumab. C-G CrCl Method was used to determine renal function. ESRD= requires hemodialysis.
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 9 | 9
participants
  Deaths | 0 | 0 | 0
  Any SAE | 3 | 5 | 7
  AEs Leading to Discontinuation | 1 | 4 | 1

4. Secondary Outcome: Number of Participants With Persistent Elotuzumab Anti-drug Antibodies (ADA) and Number of Participants ADA Positive at Cycle 2 Pre-dose.
Description: Serum samples were evaluated for the presence of ADAs using a validated bridging electrochemiluminescence (ECL) immunoassay. Samples in: Cycle 1, Day 1 0 h (pre-dose), Cycle 2, Day 1(Study Day 29), 0 h (pre-dose; 672 h post-dose), Cycle 3, Day 1, 0 h and in cycle thereafter, at end of study/discontinuation, and at 30 and 60 day follow up visits post treatment. ADA Positive Participant: baseline negative with at least one ADA positive sample at any time after initiation of treatment or baseline positive with at least one ADA positive sample at any time after initiation of treatment with a titer 9-fold greater than the baseline; Persistent Positive: ADA positive at 2 or more sequential timepoints at least 12 weeks apart; Last Sample Positive: Not persistent positive and ADA Positive Sample in the last sampling timepoint; Other Positive: not persistent positive with ADA negative sample in the last sampling; ADA Negative: no ADA positive sample after the initiation of treatment.
Time Frame: From first dose (Day 1) to last dose plus 60 days, up to Primary Endpoint (June 2014), approximately 2 years
Population: All participants with baseline ADA result and at least one on-treatment ADA result.
Measure: Number; unit: participants
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 6 | 4 | 6
participants
  Baseline ADA Positive | 1 | 0 | 0
  On-Study ADA Positive | 2 | 1 | 1
  Positive at Cycle 2 pre-dose | 2 | 0 | 1
  Persistent Positive | 0 | 0 | 0
  Last Sample Positive | 1 | 0 | 1
  Other Positive | 1 | 1 | 0
  On-Study ADA Negative | 4 | 3 | 5

5. Secondary Outcome: Number of Participants With Worst Toxicity Grade Hematology Laboratory Tests
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 was used to measure toxicity scale. Lower Limits of Normal (LLN). Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Lymphocytes absolute (abs) Gr 1: <1.5 to 0.8 *10^3 c/µL, Gr 2 <0.8 to 0.5 *10^3 c/µL, Gr 3: <0.5 to 0.2 *10^3 c/µL, Gr 4: <0.2*10^3 c/µL. Neutrophils abs: Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Leukocytes Gr 1:<LLN to 3.0 *10^3 c/µL, Gr 2; <3.0 to 2.0 *10^3 c/µL, Gr 3: <2.0 to 1.0 *10^3 c/µL, Gr 4: <1.0 *10^3 c/µL.
Time Frame: From first dose (Day 1) to last dose plus 60 days (Assessed up to July 2016, approximately 54 months)
Population: All participants who received at least one dose of study treatment (at least one dose of any drug) were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 9 | 9
participants
  Hemoglobin Any Grade | 8 | 9 | 9
  Hemoglobin Grade 3-4 | 0 | 2 | 6
  Platelet Count Any Grade | 7 | 8 | 8
  Platelet Count Grade 3-4 | 0 | 2 | 2
  Leukocytes Any Grade | 8 | 8 | 6
  Leukocytes Grade 3-4 | 3 | 1 | 2
  Lymphocytes (Abs) Any Grade | 8 | 9 | 9
  Lymphocytes (Abs) Grade 3-4 | 6 | 9 | 5
  Neutrophil Count (Abs) Any Grade | 6 | 5 | 6
  Neutrophil Count (Abs) Grade 3-4 | 3 | 1 | 2

6. Secondary Outcome: Number of Participants With Worst Toxicity Grade Renal and Liver Function Laboratory Tests
Description: NCI CTCAE, version 3.0 was used to measure toxicity scale. Lower Limits of Normal (LLN). Upper Limits of Normal (ULN). Alanine transaminase (ALT); Aspartate aminotransferase (AST); Alkaline phosphatase (ALP). ALT Grade (Gr)1:>1.0 to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. AST Gr 1: >1.0 to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Total bilirubin Gr 1: >1.0 to 1.5*ULN; Gr 2: >1.5 to 3.0*ULN; Gr 3: >3.0 to 10..0*ULN; Gr 4: >10.0.0*ULN. ALP (U/L) Gr1:>1.0 to 2.5*ULN, Gr2:>2.5 to 5.0*ULN, Gr3:>5.0 to 20.0*ULN, Gr4:>20.0*ULN. Albumin (low) Gr 1:<LLN to 3 grams per deciliter (g/dL); Gr 2: <3.0 - 2.0 g/L; Gr 3: < 2 g/dL. Creatinine Gr 1: >1 - 1.5*baseline (BL)to >ULN - 1.5*ULN; Gr 2: >1.5 - 3.0*BL to > 1.5 - 3.0*ULN; Gr 3: >3.0*BL to > 3.0 - 6.0*ULN; Gr 4: >6.0*ULN.
Time Frame: From first dose (Day 1) to last dose plus 60 days (Assessed up to July 2016, approximately 54 months)
Population: All participants who received at least one dose of study treatment (at least one dose of any drug) were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 9 | 9
participants
  ALP Any Grade | 0 | 3 | 7
  ALP Grade 3-4 | 0 | 0 | 0
  AST Any Grade | 3 | 2 | 5
  AST Grade 3-4 | 0 | 0 | 0
  ALT Any Grade | 2 | 5 | 5
  ALT Grade 3-4 | 0 | 0 | 0
  Bilirubin Any Grade | 1 | 1 | 2
  Bilirubin Grade 3-4 | 0 | 0 | 0
  Creatinine Any Grade | 0 | 9 | 9
  Creatinine Grade 3-4 | 0 | 2 | 9
  Albumin Any Grade | 2 | 7 | 7
  Albumin Grade 3-4 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Worst Toxicity Grade Chemistry Laboratory Tests
Description: Sodium high (H) Gr 1:>ULN - 150; Gr 2: >150 - 155; Gr 3: >155 - 160; Gr 4: >160 mmol/L; Sodium low(L) Gr 1:<LLN - 130; Gr 3: <130 - 120; Gr 4: <120 mmol/L. Potassium (H) Gr 1: >ULN - 5.5; Gr 2: >5.5 - 6.0; Gr 3: > 6.0 - 7.0; Gr 4: >7.0 mmol/L; Potassium (L) Gr 1: <LLN - 3.0; Gr 2: <LLN - 3.0; Gr 3: < 3.0 - 2.5; Gr 4: <2.5 mmol/L. Bicarbonate Gr1: 16-<LLN, Gr2: 11-16, Gr3, 8-11, Gr4: <8 milliequivalents per liter (mEq/L). Phosphorus Gr 1: 2.5 - <LLN, Gr2 2.0-<2.5, Gr3: 1.0-<2.0, Gr4: <1.0. Calcium (L) Gr 1: <LLN to 8.0; Gr2: 7.0 - 8.0; Gr3: 6.0-7.0; Gr 4: <6.0 mg/dL; calcium (H) Gr1:>ULN - 11.5, Gr2:>11.5 - 12.5, Gr3: 12.5 - 13.5, Gr4: >13.5.
Time Frame: From first dose (Day 1) to last dose plus 60 days (Assessed up to July 2016, approximately 54 months)
Population: All participants who received at least one dose of study treatment (at least one dose of any drug) were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 9 | 9
participants
  Sodium High Any Grade | 2 | 3 | 2
  Sodium High Grade 3-4 | 0 | 0 | 0
  Sodium Low Any Grade | 2 | 6 | 5
  Sodium Low Grade 3-4 | 1 | 1 | 0
  Potassium High Any Grade | 2 | 2 | 4
  Potassium High Grade 3-4 | 0 | 0 | 3
  Potassium Low Any Grade | 2 | 5 | 6
  Potassium Low Grade 3-4 | 0 | 2 | 1
  Bicarbonate Any Grade | 5 | 8 | 6
  Bicarbonate Grade 3-4 | 0 | 0 | 0
  Calcium High Any Grade | 1 | 0 | 3
  Calcium High Grade 3-4 | 0 | 0 | 1
  Calcium Low Any Grade | 4 | 6 | 8
  Calcium Low Grade 3-4 | 0 | 1 | 2
  Glucose High Any Grade | 7 | 9 | 7
  Glucose High Grade 3-4 | 3 | 4 | 3
  Glucose Low Any Grade | 1 | 0 | 1
  Glucose Low Grade 3-4 | 0 | 0 | 0

8. Other Pre Specified Outcome: Mean Terminal-phase Elimination Half-life (T-Half) of Elotuzumab Following Cycle 1, Day 1 Dose Administration - Grouping by Cockcroft-Gault Creatinine Clearance Method
Description: The quantification of elotuzumab in human serum was performed using validated ELISA. Cycle 1, day 1 sample times: 0 hour (h) pre-dose, end of infusion, 30 minutes (min) post end of infusion, 2 h, 4 h , and 24 h post end of infusion. Trough samples were obtained in subsequent cycles and at 30 day and 60 day follow-up visits at end of treatment. ESRD had 2 additional samples: immediately prior to and immediately after dialysis. T-Half was measured in hours (h). PK parameter renal function group assignment criteria differed slightly from the criteria for safety and efficacy analyses (specifically for the SRI group). PK criteria: All participants with at least one pretreatment value ≥ 90 mL/min were assigned to the NRF group. All those with at least one pretreatment value < 30 mL/min were assigned to the SRI group. All those with a screening diagnosis of ESRD, were assigned to the ESRD group.
Time Frame: Day 1 of Cycle 1 to 28 days post dose
Population: The analyses of PK parameters were conducted by renal functions as determined by CrCl C-G method in those participants who were treated with at least one dose of study drug and had evaluable pre- and post-treatment values.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 7 | 8
h | 204 (134.11) | 237 (107.88) | 218 (98.87)

9. Other Pre Specified Outcome: Median Time to Maximal Concentration (Tmax) of Elotuzumab Following Cycle 1, Day 1 Dose Administration - Grouping by Cockcroft-Gault Creatinine Clearance Method
Description: The quantification of elotuzumab in human serum was performed using validated ELISA. Cycle 1, day 1 sample times for all participants: 0 hour (h) pre-dose, end of infusion, 30 minutes (min) post end of infusion, 2 h, 4 h , and 24 h post end of infusion. Trough samples were obtained in subsequent cycles and at 30 day and 60 day follow-up visits at end of treatment. ESRD had 2 additional samples: immediately prior to and immediately after dialysis. Tmax was measured in hours (h). PK parameter renal function group assignment criteria differed slightly from the criteria for safety and efficacy analyses (specifically for the SRI group). PK criteria: All participants with at least one pretreatment value ≥ 90 mL/min were assigned to the NRF group. All those with at least one pretreatment value < 30 mL/min were assigned to the SRI group. All those with a screening diagnosis of ESRD, were assigned to the ESRD group.
Time Frame: Day 1 of Cycle 1 to 28 days post dose
Population: as for outcome 8
Measure: Median (Full Range); unit: h
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 7 | 8
h | 3.23 [2.9 to 4.9] | 3.87 [2.8 to 6.8] | 3.33 [2.82 to 25.92]

10. Other Pre Specified Outcome: Geometric Mean Total Body Clearance (CLT) of Elotuzumab Following Cycle 1, Day 1 Dose Administration - Grouping by Cockcroft-Gault Creatinine Clearance Method
Description: The quantification of elotuzumab in human serum was performed using validated ELISA. Cycle 1, day 1 sample times for all participants: 0 hour (h) pre-dose, end of infusion, 30 minutes (min) post end of infusion, 2 h, 4 h , and 24 h post end of infusion. Trough samples were obtained in subsequent cycles and at 30 day and 60 day follow-up visits at end of treatment. ESRD had 2 additional samples: immediately prior to and immediately after dialysis. CLT was measured in mL per hour per kilogram body weight (mL/h/kg). PK parameter renal function group assignment criteria differed slightly from the criteria for safety and efficacy analyses (specifically for the SRI group). PK criteria: All participants with at least one pretreatment value ≥ 90 mL/min were assigned to the NRF group. All those with at least one pretreatment value < 30 mL/min were assigned to the SRI group. All those with a screening diagnosis of ESRD, were assigned to the ESRD group.
Time Frame: Day 1 of Cycle 1 to 28 days post dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 7 | 8
mL/h/kg | 0.215 (46) | 0.166 (28) | 0.195 (54)

11. Other Pre Specified Outcome: Geometric Mean Apparent Volume of Distribution (Vz) of Elotuzumab Following Cycle 1, Day 1 Dose Administration - Grouping by Cockcroft-Gault Creatinine Clearance Method
Description: The quantification of elotuzumab in human serum was performed using validated ELISA. Cycle 1, day 1 sample times for all participants: 0 hour (h) pre-dose, end of infusion, 30 minutes (min) post end of infusion, 2 h, 4 h , and 24 h post end of infusion. Trough samples were obtained in subsequent cycles and at 30 day and 60 day follow-up visits at end of treatment. ESRD had 2 additional samples: immediately prior to and immediately after dialysis. Vz was measured in mL per kilogram body weight (mL/kg). PK parameter renal function group assignment criteria differed slightly from the criteria for safety and efficacy analyses (specifically for the SRI group). PK criteria: All participants with at least one pretreatment value ≥ 90 mL/min were assigned to the NRF group. All those with at least one pretreatment value < 30 mL/min were assigned to the SRI group. All those with a screening diagnosis of ESRD, were assigned to the ESRD group.
Time Frame: Day 1 of Cycle 1 to 28 days post dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Number analyzed (Participants) | 8 | 7 | 8
mL/kg | 59.4 (30) | 54.6 (20) | 61.2 (43)

ADVERSE EVENTS:
Time Frame: From first dose (Day 1) to last dose plus 60 days (Assessed up to July 2016, approximately 54 months)
Arm/Group | Elotuzumab + LD in Normal Renal Function (NRF) Participants | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants
Serious Adverse Events (participants affected / at risk) | 3/8 | 5/9 | 7/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab + LD in Normal Renal Function (NRF) Participants (N=8) | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants (N=9) | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants (N=9)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Influenza a virus test positive (Investigations) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elotuzumab + LD in Normal Renal Function (NRF) Participants (N=8) | Elotuzumab + LD in Severe Renal Impairment (SRI) Participants (N=9) | Elotuzumab + LD in End Stage Renal Disease (ESRD) Participants (N=9)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0
Scleral hyperaemia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 3 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 5
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 4
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4
Asthenia (General disorders) | 1 | 1 | 2
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Chills (General disorders) | 2 | 0 | 2
Cyst (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 6 | 4 | 7
Feeling abnormal (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 0
Infusion site bruising (General disorders) | 0 | 1 | 0
Injection site extravasation (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 3 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 4 | 4
Pain (General disorders) | 0 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 4 | 2 | 4
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Abdominal hernia infection (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 1 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 3 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2
Aspartate aminotransferase decreased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 5 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 1
Weight increased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 4 | 1
Tremor (Nervous system disorders) | 0 | 2 | 2
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Superficial vein prominence (Vascular disorders) | 0 | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.